CLINICAL TRIAL: NCT02673775
Title: Activated Macrophages and Ozone Toxicity
Brief Title: Air Pollution Study: The Effect of Ozone on the Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Howard M. Kipen, MD, MPH, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro20140001089; R01ES004738 (NIH)
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Results first posted 2023-10-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Air Pollution
Keywords: Macrophage
MeSH Terms: interventions — Environment, Controlled; Ozone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clean Air (Placebo Comparator): Subjects will be exposed to clean air for 3 hours.
  Interventions: Other: Clean Air
- Ozone (Experimental): Subjects will be exposed to 0.2 ppm ozone for 3 hours.
  Interventions: Other: Ozone

INTERVENTIONS:
Other: Clean Air — Subjects will have the clean air exposure first, followed by the ozone exposure
  Arms: Clean Air
Other: Ozone — Subjects will have the ozone exposure first, followed by the clean air exposure
  Arms: Ozone

SUMMARY:
The purpose of the study is to better understand the mechanisms of lung injury from ozone exposure. Subjects will participate in two exposure sessions: filtered air and 0.2 ppm ozone. Subjects will be asked to produce sputum through coughing after each exposure. The samples will be analyzed for macrophage activity.

DETAILED DESCRIPTION:
Subjects will be asked to come to the Rutgers EOHSI clinical center (Piscataway, NJ) for 5 study visits. A physical exam to determine eligibility will be done at the first study visit. If the subject is healthy and able to produce a sputum sample, he/she will then be scheduled for 2 3-hour exposure visits. One exposure will be to clean air and the other exposure will be to 0.2 ppm ozone. During the exposures, subjects will be requested to ride an exercise bicycle intermittently (approximately every 15 minutes). A follow-up visit for sputum collection will be scheduled either 24, 48, or 72 hours after each exposure visit. Blood, urine, and exhaled breath samples will also be collected at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women

Exclusion Criteria:

* Cardiovascular disease
* Respiratory disease
* Diabetes
* Pregnancy
* HIV infection
* History of smoking within the last 5 years
* Daily use of antioxidant supplements (e.g., Vitamin C/E, selenium, beta-carotene, lycopene, lutein, zeaxanthin, or ginkgo biloba)
* Orthopedic or rheumatological conditions that would interfere with cycle use

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard M. Kipen, MD, MPH, Principal Investigator — Rutgers School of Public Health
Locations (1):
- Environmental and Occupational Health Sciences Institute, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
The individual data will be confidential.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 135 participants from the local community were screened for eligibility between 2/1/2016 and 5/4/2022.
Pre-assignment Details: 57 were ineligible and 16 were lost to follow-up. 62 were randomized to the first exposure.
Groups:
- Ozone Exposure Was First, Followed by Clean Air Exposure: Subjects randomized to ozone first and clean air second. A washout period (at least 2 weeks) took place between exposures.
- Clean Air Exposure Was First, Followed by Ozone Exposure: Subjects randomized to clean air first and ozone second. A washout period (at least 2 weeks) took place between exposures.
Period: First Exposure
Arm/Group | Ozone Exposure Was First, Followed by Clean Air Exposure | Clean Air Exposure Was First, Followed by Ozone Exposure
Started | 25 | 37
Completed | 25 | 37
Not Completed | 0 | 0
Period: Washout (at Least 2 Weeks)
Arm/Group | Ozone Exposure Was First, Followed by Clean Air Exposure | Clean Air Exposure Was First, Followed by Ozone Exposure
Started | 25 | 37
Completed | 21 | 33
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Study paused during COVID pandemic (3/5/2020 to 9/15/2021) | 2 | 2
Period: Second Exposure
Arm/Group | Ozone Exposure Was First, Followed by Clean Air Exposure | Clean Air Exposure Was First, Followed by Ozone Exposure
Started | 21 | 33
Completed | 21 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 62 participants were randomized to a first exposure.
Groups:
- Overall: All participants who were randomized to a first exposure (N=62)
Arm/Group | Overall
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 30
  More than one race | 2
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of M1 and M2 Macrophages in the Sputum 24 Hours After Exposure.
Description: The relative concentrations of M1 and M2 macrophages in the induced sputum sample will be assessed.
Time Frame: 24 hours after exposure.
Population: The number of participants who had an adequate sputum sample collected 24 hours after each exposure.
Measure: Mean (Standard Error); unit: ratio of M2 to M1 macrophages
Arm/Group | Clean Air | Ozone
Number analyzed (Participants) | 13 | 13
ratio of M2 to M1 macrophages | 6.823 (2.413) | 1.367 (0.367)

2. Primary Outcome: Concentrations of M1 and M2 Macrophages in the Sputum 48 Hours After Exposure.
Description: The relative concentrations of M1 and M2 macrophages in the induced sputum sample will be assessed.
Time Frame: 48 hours after exposure
Population: The number of participants who had an adequate sputum sample collected 48 hours after each exposure.
Measure: Mean (Standard Error); unit: ratio of M2 to M1 macrophages
Arm/Group | Clean Air | Ozone
Number analyzed (Participants) | 9 | 9
ratio of M2 to M1 macrophages | 9.783 (3.239) | 3.449 (1.116)

3. Primary Outcome: Concentrations of M1 and M2 Macrophages in the Sputum 72 Hours After Exposure.
Description: Relative concentrations of M1 and M2 macrophages in the induced sputum sample will be assessed.
Time Frame: 72 hours after exposure.
Population: The number of participants who had an adequate sputum sample collected 72 hours after each exposure.
Measure: Mean (Standard Error); unit: ratio of M2 to M1 macrophages
Arm/Group | Clean Air | Ozone
Number analyzed (Participants) | 12 | 12
ratio of M2 to M1 macrophages | 4.623 (0.782) | 4.379 (0.623)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until the sputum sample was collected; up to 3 days after the exposure. Induced sputum was collected either 24, 48, or 72 hours after exposure; at the time of sputum collection participants were queried about any effects of the exposure including the need to see medical treatment for breathing difficulties.
Groups:
- Clean Air: Participants who received clean air exposure for 3 hours.
- Ozone: Subjects who were exposed to 0.2 ppm ozone for 3 hours.
Arm/Group | Clean Air | Ozone
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT02673775/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT02673775/SAP_001.pdf
  • Informed Consent Form (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT02673775/ICF_002.pdf